CLINICAL TRIAL: NCT07088887
Title: Bruxism Awareness as a Pre-Treatment Consideration in Dental Implantology
Brief Title: Bruxism Awareness Prior to Dental Implant Treatment
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gülbahar Ustaoğlu, associate professor, Saglik Bilimleri Universitesi
Other Study IDs: BAHAR1
Record Dates: First submitted 2025-07-11; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Bruxism
Keywords: bruxism; dental implant; Fonseca Anamnestic Index; Perceived Stress Scale-14; awareness.
MeSH Terms: conditions — Bruxism | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bruxism group: The study group included patients aged 18-65 who were systemically healthy and suitable for implant treatment. Collected data covered demographic variables (age, gender), systemic and periodontal health status, and detailed clinical findings. Bruxism was assessed both clinically-based on signs such as masseter hypertrophy and dental wear-and through self-reported questionnaires to determine its type (awake or sleep). Patients also completed the Fonseca Anamnestic Index (FAI) to evaluate temporomandibular disorder (TMD) severity and the Perceived Stress Scale-14 (PSS-14) to assess emotional stress levels. Additionally, a bruxism awareness questionnaire was administered. All evaluations were performed prior to implant surgery using standardized diagnostic forms and validated scales.
  Interventions: Other: control group

INTERVENTIONS:
Other: control group — The control group included patients aged 18-65 who were systemically healthy, had no clinical or self-reported signs of bruxism, and were eligible for implant treatment. Data collected included demographic characteristics (age, gender), systemic and periodontal health status, and clinical examination findings confirming the absence of bruxism. These patients also completed the Fonseca Anamnestic Index (FAI) to assess temporomandibular disorder (TMD) symptoms and the Perceived Stress Scale-14 (PSS-14) to evaluate emotional stress levels. A bruxism awareness questionnaire was also applied to determine baseline knowledge in individuals without bruxism. All assessments were conducted before implant surgery using standardized diagnostic tools.

SUMMARY:
Bruxism is a parafunctional habit characterized by clenching or grinding of the teeth and/or mandibular thrusting, which may occur during sleep or wakefulness. It is associated with various dental complications, including implant failures. Despite its prevalence, awareness of bruxism among patients remains limited, and diagnostic methods vary. This study aims to evaluate the presence and type of bruxism in patients undergoing dental implant treatment and to assess their awareness levels. The findings may help prevent implant-related complications by supporting early identification and appropriate management of bruxism.

Research Questions What is the prevalence of awake and sleep bruxism in patients scheduled for dental implant treatment?

To what extent are patients aware of their bruxism habits prior to treatment?

What are the most common signs and symptoms of bruxism observed in this patient group?

Is there a correlation between patients' self-reported bruxism and clinical findings?

Can increased bruxism awareness before implant procedures help reduce the risk of future implant and prosthetic complications?

DETAILED DESCRIPTION:
This observational study involves systemically healthy adult patients scheduled for dental implant treatment at a university dental faculty. Clinical examinations were performed to detect characteristic signs of bruxism, and validated self-report tools-including the Bruxism Questionnaire, Fonseca Anamnestic Index, and Perceived Stress Scale-were used to assess both subjective awareness and emotional stress. Additionally, a customized awareness questionnaire was administered to evaluate patients' perceptions and knowledge of bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Participants included in the study were individuals aged between 18 and 65 years,
* who were systemically healthy and
* able to comprehend and respond to the questionnaire items

Exclusion Criteria:

* Individuals with intellectual disabilities,
* suicidal tendencies, dementia,
* or psychosis were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of 150 systemically healthy adult patients aged 18 to 65 who applied to the Department of Periodontology at Gülhane Faculty of Dentistry, University of Health Sciences, Ankara, Turkey, between March and June 2025. All participants were seeking dental implant therapy. The sample represents a clinical population attending a tertiary care academic dental center, with diverse educational and socioeconomic backgrounds. Patients with intellectual disabilities, psychiatric disorders, or conditions impairing questionnaire comprehension were excluded. This observational cohort was selected to evaluate the presence of bruxism and patient awareness prior to implant placement.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
diagnosis of bruxism | Baseline (before dental implant surgery)
  Bruxism assessment in this study was based on both clinical examination and self-reported measures. Clinical diagnosis followed the 2018 international consensus criteria, requiring at least two of the following signs: masseter muscle pain or hypertrophy (extraoral), dental wear, linea alba on the buccal mucosa, or recurrent restoration failures (intraoral). Self-reported bruxism was evaluated using a standardized questionnaire based on Lobbezoo et al.'s grading system, distinguishing between awake and sleep bruxism.

SECONDARY OUTCOMES:
Stress Level | Baseline (before dental implant surgery)
  The Perceived Stress Scale-14 (PSS-14), developed by Cohen et al. in 1983, was used to assess the level of emotional stress. This self-reported questionnaire comprises 14 items that evaluate the frequency of stress-related thoughts and feelings experienced by the respondent over the past month. Participants rate each item on a four-point Likert scale ranging from "never" to "very often." The total score ranges from 0 to 56, with higher scores indicating greater levels of perceived emotional stress.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLBAHAR USTAOĞLU, Assoc Prof, Principal Investigator — GÜLHANE DİŞ HEKİMLİĞİ FAKÜLTESİ
Locations (1):
- Health Sciences University Gulhane Faculty of Dentistry,, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No